CLINICAL TRIAL: NCT00447343
Title: Mapping of the Sensorimotor Cortex in Cervical Myelopathy Using Functional Magnetic Resonance Imaging and Magnetic Resonance Spectroscopy
Brief Title: Reorganization of Brain Functions in Patients With Cervical Myelopathy Using fMRI and MRS
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); American Association of Neurological Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: R-04-022; 09994
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Diseases
Keywords: Functional MRI; Cervical myelopathy; Cervical radiculopathy; Brain plasticity and regeneration
MeSH Terms: conditions — Spinal Cord Diseases; Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment group: Patients with cervical myelopathy undergoing decompressive cervical spine surgery will have two scans (pre-operatively and 6 months post-operatively).
  A blinded investigator will administer questionnaires at each time point.
  Interventions: Procedure: Decompressive cervical spine surgery; Procedure: fMRI and MRS scan
- Control group: Healthy Volunteers will have two scans 6 months apart.
  A blinded investigator will administer questionnaires at each time point.
  Interventions: Procedure: fMRI and MRS scan

INTERVENTIONS:
Procedure: Decompressive cervical spine surgery — Treatment group (25 patients) will undergo decompressive anterior cervical spine surgery
  Healthy volunteers will ONLY undergo two scans 6 months apart.
  Groups: Treatment group
Procedure: fMRI and MRS scan — A scan pre-op and 6 months post-op.

SUMMARY:
Decompressive surgery to relieve symptoms of spinal cord compression due to dysfunction, such as arthritis, has proved variable in success. Past research has reported that approximately one-third of surgery patients improved, one-third remained the same and one-third worsened. Currently, there are no reliable tests that can predict the outcome following surgery. We are hoping that this study will change that.

Using functional MRI (fMRI), we wish to investigate the relationship between clinical symptoms and the recovery of brain activation following surgery. One can also track the concentrations of different chemicals (metabolites) by using magnetic resonance spectroscopy (MRS). We hypothesize that the recovery of normal brain activation patterns will coincide with clinical improvement. Our objective in this study is to explore the potential role of fMRI as a tool to prognose patients with cervical myelopathy.

Twenty-five patients with cervical myelopathy will be imaged using a high-powered (3 Tesla) fMRI scanner before and six months following surgery. In addition, ten healthy controls will be imaged to provide a baseline measure. Both the patient and control groups will complete questionnaires at the time of their scans. These will provide information concerning the subjective experience of the individuals throughout recovery. We will compare brain activation patterns of control and patient groups to investigate how the brain heals following decompressive surgery.

DETAILED DESCRIPTION:
Degenerative arthritis is a universal concomitant of human aging, affecting 51% of the adult population. Arthritis of the spine is the most common cause of acquired spinal cord dysfunction and can manifest in subtle symptoms, such as diminished balance and dexterity, or profound symptoms, such as paralysis and incontinence. In cases where dysfunction results in severe spinal cord compression, surgery is performed. However, surgical outcomes are not always beneficial. Past research has reported that approximately one-third of surgery patients improved, one-third remained the same and one-third worsened. Currently, there are no reliable tests that can predict outcome following surgery. We are hoping that this study will change that.

Twenty-five patients will undergo 45 minute imaging sessions pre-operatively and six months post-operatively. Ten controls will undergo 45 minute imaging sessions twice to provide a baseline comparison and reproducibility. During each session, one motor task (finger tapping) and 1 sensory task (hand brushing) will be performed for 2 minutes at 10 second intervals. We wish to compare the change in volume extent, and location, and intensity of brain activation levels before and after surgery. We will also compare fMRI signal response differences between controls and patients. We hypothesize that the degree to which brain activation shifts towards normalcy (that of controls) will correlate with the degree of neurological recovery postoperatively.

Data will be analyzed using software developed at the Robarts Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* All Participants will be

  1. between 18 and 75 years of age
  2. right handed
  3. with normal/corrected hearing and vision
  4. native speakers of Canadian or American English
  5. must be competent to give consent.
* Cervical Myelopathy Patients will be:

  1. Undergoing a first time cervical decompression for cervical spondylosis causing myelopathy secondary to spinal cord compression which is documented by a diagnostic procedure ( CT and/or MRI ).
  2. Spinal cord compression from the cervicomedullary junction to the C7-T1 disc level.
  3. Ability and willingness to participate in a follow-up fMRI study at 6 months following surgery.
* Healthy Control Volunteers will be:

  1. Volunteers from the Dept. of Clinical Neurological Sciences

Exclusion Criteria:

* Cervical Myelopathy Patients must not:

  1. have any pre-existing medical conditions (e.g. significant renal or hepatic disease)
* Healthy control volunteers must not:

  1. have a pre-existing diagnosis or history of a neurological disorder.
* All participants must not:

  1. have any potential magnetic metal fragments in their body except for titanium implants placed at the time of surgery will be excluded. Dental work is non-magnetic and does not require participant exclusion.
* Participants who fall into the following categories will not be tested in the 4T scanner:

  1. claustrophobia
  2. pacemaker or other electronic implants
  3. being a welder or soldier
  4. having been injured by a metallic object that was not removed
  5. being pregnant or trying to conceive
  6. women of childbearing potential who are not using an effective method of contraception
  7. cerebral aneurysm clips.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-five patients and ten controls will be recruited from the Clinical Neurological Sciences outpatient clinic at the London Health Sciences Centre, University Campus
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Measure the volume of activation and signal intensity using fMRI and MRS. | 2 scans 6 months apart

SECONDARY OUTCOMES:
Clinical changes will be measured using validated disease specific scoring instruments including the Japanese Orthopedic Association scale (JOA), Nurick, ASIA/ISCOS Impairment Scale, Short Form Health Survey (SF-36) and the Neck Disability Index (NDI). | 2 scans 6 months apart

CONTACTS AND LOCATIONS:
Overall Officials: Neil Duggal, M.D., M.Sc., Principal Investigator — London Health Sciences Center; Robert Bartha, Ph.D, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Background] BRAIN WR, NORTHFIELD D, WILKINSON M. The neurological manifestations of cervical spondylosis. Brain. 1952 Jun;75(2):187-225. doi: 10.1093/brain/75.2.187. No abstract available. PMID 14934989
- [Background] Bunge RP, Puckett WR, Becerra JL, Marcillo A, Quencer RM. Observations on the pathology of human spinal cord injury. A review and classification of 22 new cases with details from a case of chronic cord compression with extensive focal demyelination. Adv Neurol. 1993;59:75-89. No abstract available. PMID 8420126
- [Background] Carol MP, Ducker TB. Cervical spondylitic myelopathies: surgical treatment. J Spinal Disord. 1988;1(1):59-65. PMID 2980063
- [Background] Curt A, Alkadhi H, Crelier GR, Boendermaker SH, Hepp-Reymond MC, Kollias SS. Changes of non-affected upper limb cortical representation in paraplegic patients as assessed by fMRI. Brain. 2002 Nov;125(Pt 11):2567-78. doi: 10.1093/brain/awf250. PMID 12390981
- [Background] Hunt WE. Cervical spondylosis: natural history and rare indications for surgical decompression. Clin Neurosurg. 1980;27:466-80. doi: 10.1093/neurosurgery/27.cn_suppl_1.466. PMID 7273568
- [Background] LaRocca H. Cervical spondylotic myelopathy: natural history. Spine (Phila Pa 1976). 1988 Jul;13(7):854-5. doi: 10.1097/00007632-198807000-00028. No abstract available. PMID 3057650
- [Background] Lunsford LD, Bissonette DJ, Jannetta PJ, Sheptak PE, Zorub DS. Anterior surgery for cervical disc disease. Part 1: Treatment of lateral cervical disc herniation in 253 cases. J Neurosurg. 1980 Jul;53(1):1-11. doi: 10.3171/jns.1980.53.1.0001. PMID 7411195
- [Background] Morio Y, Teshima R, Nagashima H, Nawata K, Yamasaki D, Nanjo Y. Correlation between operative outcomes of cervical compression myelopathy and mri of the spinal cord. Spine (Phila Pa 1976). 2001 Jun 1;26(11):1238-45. doi: 10.1097/00007632-200106010-00012. PMID 11389390
- [Background] Rowland LP. Surgical treatment of cervical spondylotic myelopathy: time for a controlled trial. Neurology. 1992 Jan;42(1):5-13. doi: 10.1212/wnl.42.1.5. PMID 1734322
- [Background] Teramoto T, Ohmori K, Takatsu T, Inoue H, Ishida Y, Suzuki K. Long-term results of the anterior cervical spondylodesis. Neurosurgery. 1994 Jul;35(1):64-8. doi: 10.1227/00006123-199407000-00010. PMID 7936154
- [Background] Yonenobu K, Hosono N, Iwasaki M, Asano M, Ono K. Laminoplasty versus subtotal corpectomy. A comparative study of results in multisegmental cervical spondylotic myelopathy. Spine (Phila Pa 1976). 1992 Nov;17(11):1281-4. PMID 1462201